CLINICAL TRIAL: NCT02152306
Title: A Randomized, Double-blind Multicenter, Phase III Study to Evaluate the Efficacy and Safety of Combination of Fimasartan/Amlodipine Versus Fimasartan Monotherapy in Patients With Essential Hypertension Who Fail to Respond Adequately to Fimasartan Monotherapy.
Brief Title: Fimasartan/Amlodipine Combination Phase III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Gachon University Gil Medical Center (Other); The Catholic University of Korea (Other); Kangbuk Samsung Hospital (Other); Kyungpook National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Korea University Guro Hospital (Other); Korea University Anam Hospital (Other); DongGuk University (Other); Dong-A University Hospital (Other); Pusan National University Hospital (Other); Seoul National University Bundang Hospital (Other); Seoul National University Hospital (Other); Asan Medical Center (Other); Pusan National University Yangsan Hospital (Other); Wonju Severance Christian Hospital (Other); Gangnam Severance Hospital (Other); Severance Hospital (Other); Ulsan University Hospital (Other); Inje University (Other); Inje University Haeundae Paik Hospital (Other); Chonnam National University Hospital (Other); Jeju National University Hospital (Other); Chungnam National University (Other); Hanyang University Seoul Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FAC-CT-301
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; Fimasartan and Amlodipine; Antihypertension
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fimasartan and Amlodipine (Experimental): Combination of Fimasartan and Amlodipine
  Interventions: Drug: Fimasartan and Amlodipine
- Fimasartan (Active Comparator): Fimasartan Monotherapy
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan and Amlodipine
  Arms: Fimasartan and Amlodipine
Drug: Fimasartan
  Arms: Fimasartan

SUMMARY:
The aim of this study is to ensure the superiority of Fimasartan/Amlodipine combination in hypotensive effect after 8 weeks of treatment over Fimasartan monotherapy in patients with hypertension who have no response to Fimasartan 60mg monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily signed informed consent for participating in this clinical trial
2. Male and Female between 20 and 75 years old
3. Patients with essential hypertension
4. Patients who is unresponsive to Fimasartan 60mg monotherapy for 4 weeks (i.e. the mean SiDBP from 3 times of measurement is 140mmHg ≤ SiSBP <180 mmHg)
5. Understand the trial procedures and be willing to cooperate and complete the trial.

Exclusion Criteria:

1. Severe Hypertension patients (SiDBP ≥ 110mmHg and/or SiSBP ≥ 180mmHg)
2. Subjects with the difference between blood pressures from a selected arm, SiDBP ≥10 mmHg or SiSBP ≥20 mmHg, at screening assessment
3. Secondary hypertension patients, but not limited to the following disease;(example: renovascular disease, adrenal medullary and cortical hyperfunctions, coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromo-cytoma, polycystic kidney disease, etc.)
4. Clinically significant renal function abnormality in the laboratory results at screening (i.e. serum creatine ≥ 1.5 times upper normal limit (UNL)), liver function abnormality (ALT, AST ≥ 2 times upper normal limit (UNL)), severe fatty liver disease that requires medication
5. Clinically significant Hypokalemia(Less than 3.5mmol/L), Hyperkalemia(exceeded 5.5mmol/L)
6. Subjects with following surgical and internal disease that may affect absorption, distribution, metabolism or excretion of drugs and have conditions which include the following (but are not limited to): history of major gastrointestinal surgeries including gastrectomy, gastro-enterostomy or bowel resection, gastrointestinal bypass graft and stapling; current active gastritis, ulcer, gastrointestinal and rectal bleeding, presence of active inflammatory bowel syndrome within the past 12 months; or clinically significant urinary obstruction at discretion of investigator
7. Subjects with depletion of body fluid or sodium ion not able to correct
8. Subjects with severe insulin-dependent Diabetes Mellitus (DM) or chronic DM (HbA1c>9%, dosage of an oral hypoglycemic agent was modified within the past 12 weeks, or use of active insulin treatment at screening)
9. Subjects with severe heart disease (heart failure New York Heart Association(NYHA) Class III and IV), or history of any of the followings within the past 6 months; ischemic heart disease(e.g. angina pectoris, myocardial infarction), peripheral vascular disease, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft.
10. Subjects with clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or any other clinical significant arrhythmia conditions at discretion of investigator.
11. Subjects with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve stenosis, or mitral valve stenosis.
12. Subjects with severe cerebrovascular disorder (e.g. stroke, cerebral infarction or cerebral hemorrhage within the past 6 months).
13. Subjects with chronic inflammatory disease requiring an chronic anti-inflammatory therapy, Past or current medical history with wasting disease, autoimmune diseases (e.g. rheumatoid arthritis, systemic lupus erythematosus ) or connective tissue disease.
14. Subjects with known moderate or malignant retinosis (e.g. retinal hemorrhage, visual disturbance or retinal microaneurysm in the past 6 months).
15. Subjects with hepatitis B (including positive test for HBsAg), hepatitis C-positive.
16. Subjects with history or evidence of abusing drugs or alcohol within the past 2 years.
17. Medical history with hypersensitivity to angiotensin II antagonist-based drugs or calcium-channel blockers
18. Subjects with hereditary disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
19. Pregnant women and lactating female
20. Women of childbearing potential who are not using effective contraceptive methods. (Excluding subjects who had surgically sterilized. All women of childbearing potential who did not have surgical sterilization must prove negative in a pregnancy test, and continue to use accepted and effective contraceptive methods until the end of the study in order to participate. Not accepted contraceptive method: Periodic abstinence and celibacy (e.g. Basic body temperature method, menstrual cycle calculation), hormonal contraceptives.
21. Subject who is participating in another trial or took other investigational product within12 weeks from the screening visit
22. Medical history of all kinds of malignant tumor including leukemia and lymphoma in the past 5 years
23. A subject with other reasons not specified above that, ineligible to participate in this clinical trial at discretion of study investigators.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change of Sitting Systolic Blood Pressure(SiSBP) at week 8 of Investigational Product(IP) Administration from the Baseline | 8 weeks from Baseline Visit
  To compare the difference of Mean Systolic Blood Pressure at 8 weeks from baseline visit

SECONDARY OUTCOMES:
Change of Sitting Systolic Blood Pressure(SiSBP) at week 4 of Investigational Product(IP) Administration from the Baseline | 4 weeks from Baseline Visit
Changes of Sitting Diastolic Blood Pressure(SiDBP) at week 4 and 8 of Investigational Product(IP) Administration from the Baseline | 4 and 8 weeks from Baseline Visit
Response rate of the Blood Pressure at week 8 of Investigational Product(IP) Administration | 8 weeks from Baseline Visit
The Normalization ratio of Blood Pressure at week 8 of Investigational Product(IP) Administration | 8 weeks from Baseline Visit

OTHER OUTCOMES:
Adverse Events | 12 weeks from Screening Visit
Adverse Changes in Laboratory Test Results | 12 weeks from Screening Visit
Adverse Changes in Electrocardiography (ECG) | 12 weeks from Screening Visit

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Ho Kim, Ph.D., Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Bundang, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim KI, Shin MS, Ihm SH, Youn HJ, Sung KC, Chae SC, Nam CW, Seo HS, Park SM, Rhee MY, Kim MH, Cha KS, Kim YJ, Kim JJ, Chun KJ, Yoo BS, Park S, Shin ES, Kim DS, Il Kim D, Kim KH, Joo SJ, Jeong JO, Shin J, Kim CH. A Randomized, Double-blind, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of Fimasartan/Amlodipine Combined Therapy Versus Fimasartan Monotherapy in Patients With Essential Hypertension Unresponsive to Fimasartan Monotherapy. Clin Ther. 2016 Oct;38(10):2159-2170. doi: 10.1016/j.clinthera.2016.07.008. Epub 2016 Aug 5. PMID 27502326